CLINICAL TRIAL: NCT00896012
Title: Phase 4 Study: Comparison of Myfortic and Early Rapamycin Conversion vs. Low-Dose Tacrolimus in Preventing Acute Rejection and Chronic Allograft Fibrosis: A Protocol Biopsy Directed Approach
Brief Title: Kidney Biopsy Controlled Trial of Calcineurin Inhibitor Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Novartis (Industry); University of Washington (Other)
Responsible Party: Principal Investigator, Oleh Pankewycz, MD, Nephrology, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AUS59
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplant; Immunosuppression drugs; Rapamune; tacrolimus; calcineurin inhibitor; Kidney Biopsy, Needle
MeSH Terms: interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Low-dose tacrolimus arm (Experimental): Patients in this group will continue to receive tacrolimus at reduced doses. Doses will be titrated to achieve tacrolimus trough blood levels between 4 and 6. Myfortic at doses of 720 mg BID and steroids will be continued for the duration of the study (12 months). All patients will undergo a second protocol biopsy at 12 months.
  Interventions: Procedure: Kidney Biopsy; Drug: Tacrolimus
- 2. Rapamune conversion arm: (Experimental): Patients in this group will undergo a gradual conversion from tacrolimus to Rapamune therapy. Tacrolimus will be withdrawn progressively over a period of 7-10 days. Dosage adjustments will be made with the aim of reducing the blood levels of tacrolimus by 25% every other day until tacrolimus is discontinued. Rapamune will be given at a dose of 5mg/day for two days beginning at the initiation of tacrolimus reduction. Thereafter, Rapamune will be given at a dose of 3 mg/day. The dose of Rapamune will be titrated to achieve a blood level (by HPLC) between 5 and 10 for the duration of the study.
  Interventions: Procedure: Kidney Biopsy; Drug: Rapamune (sirolimus/rapamycin)

INTERVENTIONS:
Procedure: Kidney Biopsy — Skin over the kidney will be cleansed and disinfected. The skin and deeper tissue will be numbed with novocaine like solution. A special needle will be inserted guided by ultrasound into the kidney for an instant to withdraw the small specimen.
Drug: Rapamune (sirolimus/rapamycin) — Rapamune will be given at a dose of 5mg/day for two days beginning at the initiation of tacrolimus reduction. Thereafter, Rapamune will be given at a dose of 3 mg/day. The dose of Rapamune will be titrated to achieve a blood level (by HPLC) between 5 and 10 for the duration of the study.
  Arms: 2. Rapamune conversion arm:
Drug: Tacrolimus — Patients in this group will continue to receive tacrolimus at reduced doses. Doses will be titrated to achieve tacrolimus trough blood levels between 4 and 6. Myfortic at doses of 720 mg BID and steroids will be continued for the duration of the study (12 months).
  Arms: 1. Low-dose tacrolimus arm

SUMMARY:
Current therapy to prevent organ rejection relies on the use of calcineurin inhibitors either cyclosporine or tacrolimus. Although these agents have been very successful in preventing early acute rejection, this success has not translated into improved long-term kidney transplant function. One of the important factors that leads to premature kidney transplant failure is chronic allograft nephropathy (CAN). CAN is characterized by progressive interstitial fibrosis or "scarring", vascular wall thickening, and finally glomerular sclerosis leading to slow progressive loss of kidney function. Calcineurin inhibitors have been shown to play an important role in the pathogens of CAN. Renal transplant recipients in whom calcineurin inhibitors are discontinued enjoy better and longer kidney function. Therefore, immunosuppressive strategies are being designed with the intention of withdrawing calcineurin inhibitors.

The purpose of this trial is to test if tacrolimus can be safely substituted by sirolimus (Rapamycin) and this substitution will yield improved renal function, less CAN and better graft survival rates over the first year.

DETAILED DESCRIPTION:
The purpose of this study is to determine if tacrolimus can be safely lowered to potentially non-nephrotoxic levels or discontinued completely in favor of Rapamycin 3 months after kidney transplantation. In this study, all patients will be maintained on full-dose (720 mg BID) mycophenolate sodium (Myfortic) to ensure adequate immunosuppression. In addition, we will compare the immunosuppressive regimens of Rapamune/mycophenolate sodium/Prednisone to Low-Dose Prograf/ mycophenolate sodium /Prednisone for their long-term effects on renal function, cardiovascular risk factors, subclinical rejection and chronic allograft fibrosis.

We also plan to examine the clinical benefit of protocol biopsies. The first protocol biopsy would occur at the time of implantation. This would provide an assessment of the state of the donor kidney. The severity of donor disease would provide a baseline to which all subsequent biopsies can be compared. The second protocol biopsy would be performed at the time of tacrolimus withdrawal. Patients found to have subclinical rejection on this biopsy would not undergo tacrolimus withdrawal but may benefit from increased immunosuppression. The protocol biopsy would provide an additional level of safety ensuring that only "low-risk" (histologically) patients undergo tacrolimus withdrawal. A third biopsy would be performed one year after transplantation. Renal allograft tissue would be examined for the presence of progressive fibrosis or persistent subclinical rejection both of which lead to graft failure. The efficacy of tacrolimus withdrawal can be assessed using both clinical and pathologic criteria.

A third aim of this trial is to examine whether changes in immunosuppressive therapy leads to differential expression of immunological markers or serum mediators such as cytokines. Recent studies suggest that, in vitro, thymoglobulin induces the generation of "regulatory" cells. This study will examine the in vivo relevance of this novel observation. In addition, we will measure the circulatory mediators of renal fibrosis to examine if the two treatment arms differ in their effects on such cytokine/growth factors. Blood samples will be collected and the PBMC will be analyzed by FACS for their composition and the presence of cell surface antigens that may reflect a state of immunological regulation or "suppression". Tissue samples will be analyzed by immunohistochemistry for the presence of immunologically relevant cellular subtypes such as CD4/CD25 regulatory T cells. Serum samples will be collected and analyzed for cytokine or growth factor expression.

ELIGIBILITY:
Inclusion Criteria:

1. All patients receiving their first renal allograft transplant will be considered eligible for study
2. Patients receiving both living and cadaveric donors will be eligible

Exclusion Criteria:

1. If less than 18 years of age
2. Severe hyperlipidemia
3. If pregnant or cannot comply with proper birth control during the study
4. Recipients of kidney together with another solid organ or bone marrow transplant
5. Patients receiving any investigational medications or participating in a clinical trial
6. Patients receiving a second or third renal allograft
7. PRA > 30%
8. Active infections
9. Chronic antiarrhythmic therapy for ventricular arrhythmia
10. Malignancy except for basal cell carcinoma
11. HIV
12. ANC count < 1,000/ mm3, Platelet count < 100,00/mm3
13. Fasting triglycerides > 400 mg/dl and cholesterol > 300 mg/dl
14. HCV-positive, HBVSAg-positive, HBVCoreAb-positive and HBVSAntibody negative or HCV/HBV co-infected patients
15. Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Laftavi, MD, FACS, Principal Investigator — University at Buffalo School of Medicine Deparment of Surgery; Oleh G. Pankewycz, MD, Principal Investigator — University at Buffalo
Locations (1):
- Buffalo General Hospital Multi-Organ Transplant Department, Buffalo, New York, United States

REFERENCES:
- [Background] Oberbauer R, Kreis H, Johnson RW, Mota A, Claesson K, Ruiz JC, Wilczek H, Jamieson N, Henriques AC, Paczek L, Chapman J, Burke JT; Rapamune Maintenance Regimen Study Group. Long-term improvement in renal function with sirolimus after early cyclosporine withdrawal in renal transplant recipients: 2-year results of the Rapamune Maintenance Regimen Study. Transplantation. 2003 Jul 27;76(2):364-70. doi: 10.1097/01.TP.0000074360.62032.39. PMID 12883194
- [Background] Ruiz JC, Campistol JM, Grinyo JM, Mota A, Prats D, Gutierrez JA, Henriques AC, Pinto JR, Garcia J, Morales JM, Gomez JM, Arias M. Early cyclosporine a withdrawal in kidney-transplant recipients receiving sirolimus prevents progression of chronic pathologic allograft lesions. Transplantation. 2004 Nov 15;78(9):1312-8. doi: 10.1097/01.tp.0000137322.65953.0a. PMID 15548969
- [Background] Mota A, Arias M, Taskinen EI, Paavonen T, Brault Y, Legendre C, Claesson K, Castagneto M, Campistol JM, Hutchison B, Burke JT, Yilmaz S, Hayry P, Neylan JF; Rapamune Maintenance Regimen Trial. Sirolimus-based therapy following early cyclosporine withdrawal provides significantly improved renal histology and function at 3 years. Am J Transplant. 2004 Jun;4(6):953-61. doi: 10.1111/j.1600-6143.2004.00446.x. PMID 15147430
- [Background] Larson TS, Dean PG, Stegall MD, Griffin MD, Textor SC, Schwab TR, Gloor JM, Cosio FG, Lund WJ, Kremers WK, Nyberg SL, Ishitani MB, Prieto M, Velosa JA. Complete avoidance of calcineurin inhibitors in renal transplantation: a randomized trial comparing sirolimus and tacrolimus. Am J Transplant. 2006 Mar;6(3):514-22. doi: 10.1111/j.1600-6143.2005.01177.x. PMID 16468960
- [Background] Salvadori M, Holzer H, de Mattos A, Sollinger H, Arns W, Oppenheimer F, Maca J, Hall M; ERL B301 Study Groups. Enteric-coated mycophenolate sodium is therapeutically equivalent to mycophenolate mofetil in de novo renal transplant patients. Am J Transplant. 2004 Feb;4(2):231-6. doi: 10.1046/j.1600-6143.2003.00337.x. PMID 14974944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants who received their first kidney transplant were eligible to participate. Recruitment occurred from January 2008 until October 2010.
Pre-assignment Details: Of the total 58 participants enrolled in the study, 6 participants were not randomized to either the Low Dose Tacrolimus or Rapamycin Conversion arm. Only those showing no evidence of subclinical rejection or borderline changes on 3-month protocol biopsy were eligible for randomization.
Period: Overall Study
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm:
Started | 29 | 23
Completed | 18 | 12
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm: | Total
Number analyzed (Participants) | 29 | 23 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.4) | 51.1 (13.6) | 54.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 21 | 15 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 1 | 0 | 1
  Race/Ethnicity: Asian | 0 | 1 | 1
  Race/Ethnicity: Black or African American | 4 | 3 | 7
  Race/Ethnicity: White | 22 | 16 | 38
  Race/Ethnicity: Hispanic or Latino | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 23 | 52
Donor Type [Count of Participants; unit: Participants]
  Living Donor | 13 | 15 | 28
  Deceased Donor | 16 | 8 | 24
Diagnosis [Count of Participants; unit: Participants]
  Diabetes | 16 | 7 | 23
  Hypertension | 6 | 3 | 9
  Other/Unknown | 7 | 13 | 20
Post-kidney transplant function [Count of Participants; unit: Participants]
  Delayed graft function | 5 | 1 | 6
  Immediate graft function | 24 | 22 | 46
Donor type-Expanded criteria donors [Count of Participants; unit: Participants]
  Expanded criteria donors | 7 | 1 | 8
  Non-expanded criteria donors | 22 | 22 | 44
Total rATG dose [Mean (Standard Deviation); unit: mg/kg] | 2.9 (.79) | 3.0 (.32) | 3.0 (.63)
HLA mismatch [Mean (Standard Deviation); unit: mismatched antigens] | 3.7 (1.7) | 3.8 (1.4) | 3.8 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Survival at 12 Months
Description: Graft survival is defined as no rejection or inflammation at 12 months.
Time Frame: Number of participants biopsied at 12 months post-transplant
Population: At 12 month, patients underwent a second surveillance biopsy. All biopsies were reviewed and scored using the 2005 updated Banff 1997 criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm:
Number analyzed (Participants) | 29 | 23
Participants | 18 | 12

2. Primary Outcome: Either Equivalent or Improved Estimated Glomerular Filtration Rate (eGFR) at One Year in the Rapamycin Group
Description: Estimated glomerular filtration rate (eGFR) was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
Time Frame: 1 year post-transplant
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm:
Number analyzed (Participants) | 29 | 23
mL/min
  eGFR at 1 Month | 65.5 (16.8) | 58.3 (13.6)
  eGFR at 3 Months | 68.6 (18.1) | 58.7 (13.7)
  eGRF at 6 Months | 75 (19) | 67 (14)
  eGRF at 12 Months | 74 (15) | 66 (18)
Statistical Analysis 1: Comparison: 1. Low-dose Tacrolimus Arm vs 2. Rapamune Conversion Arm:; Statistical analysis was performed by analysis of variance and Student t test for estimated glomerular filtration rate (eGFR) at 12 months. Chi-square analysis was used for demographics data; Test type: Other; p = 0.222, t-test, 2 sided — Significance was considered to be P < .05

3. Primary Outcome: Improved Histology at 12 Months in the Rapamycin Group
Description: Chronic allograft damage index (CADI) scores. It's a sum score of six histo- pathological lesions commonly seen in biopsies taken from transplanted kidneys that correlate with the function and outcome of the graft. The maximum CADI score can go up to 18. In this case the lesions found were Interstitial fibrosis (IF) and Tubular Atrophy (TA) subscales from 0 (min) to 5 (max) . A score of 0 to 1 means absence of chronic allograft damage, a score of 4 is severe damage. .
Time Frame: 3 and 12 months
Population: At one year the number of participants in LowTAC group was n=18 and Sirolimus group n= 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm:
Number analyzed (Participants) | 29 | 23
score on a scale
  CADI Score at 3-Month Randomization Follow-Up | 1.1 (1.3) | 1.0 (1.5)
  CADI Score at 12-Month Randomization Follow-up: number analyzed (Participants) | 18 | 12
  CADI Score at 12-Month Randomization Follow-up | 2.8 (2.4) | 2.0 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse Event data collection occurred from Transplant Day 0 to 12 months post-transplant.
Arm/Group | 1. Low-dose Tacrolimus Arm | 2. Rapamune Conversion Arm:
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/29 | 6/23
Other Adverse Events (participants affected / at risk) | 10/29 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1. Low-dose Tacrolimus Arm (N=29) | 2. Rapamune Conversion Arm: (N=23)
Chest Pain (Cardiac disorders) | 1 | 0
Elevated Creatinine (Renal and urinary disorders) | 2 | 0
Fever (Infections and infestations) | 0 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Humoral Kidney Transplant Rejection (Renal and urinary disorders) | 0 | 1
Atrial Arrhythmia (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic Foot Infection (Infections and infestations) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Motor Vehicle Accident (Social circumstances) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Prostate Cancer (Reproductive system and breast disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Ventral Hernia Repair (Surgical and medical procedures) | 1 | 0
Non-Cardiac Chest Pain (Reproductive system and breast disorders) | 1 | 0
Acute Cellular Kidney Rejection (Renal and urinary disorders) | 0 | 1
Pancreas Transplant (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1. Low-dose Tacrolimus Arm (N=29) | 2. Rapamune Conversion Arm: (N=23)
Bacterial Infection (Infections and infestations) | 0 | 6
Leukopenia (Blood and lymphatic system disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3
BK Infection (Infections and infestations) | 0 | 3
Fever (Infections and infestations) | 2 | 0
Sinus Infection (Infections and infestations) | 0 | 2
Toe Infection (Infections and infestations) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No